CLINICAL TRIAL: NCT06942338
Title: Comparative Evaluation of Body Temperature Measurement Using the CardioWatch 2870-2 and Invasive Temperature Monitoring in an Intensive Care Setting.
Brief Title: Comparative Evaluation of Body Temperature Measurement Using the CardioWatch 287-2 in an Intensive Care Setting.
Acronym: ICU-temp
Status: Not yet recruiting | Type: Observational
Sponsor: Corsano Health B.V. (Industry)
Responsible Party: Sponsor
Other Study IDs: ICU-temp
Record Dates: First submitted 2025-04-09; First posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: ICU Hospitalization; Surgical Intervention
Keywords: wristband; wearable; body temperature; validation; rectal temperature; remote monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Patients admitted to the ICU or recovery room with and without fever: We aim to include 120 individuals (mixed gender), of which 30-50% are displaying fever (>38°C), who are administered to the intensive care unit or the recovery room of the Reinier de Graaf Gasthuis.
  Interventions: Device: Corsano CardioWatch 287-2

INTERVENTIONS:
Device: Corsano CardioWatch 287-2 — Temperature readings from wearable Cardiowatch BT sensor, wearable Radius-T BT sensor, tympanic temperature and rectal temperature will be collected. Each participant will remain in the study as long as the rectal temperature is measured with a maximum of 24 hours. Other than the wearable Cardiowatch, the Radius-T sensors, and the rectal thermometer no additional interventions will take place due to the study. Temperature monitoring of patients will be performed according to hospitals routine care and will not be affected by the study. Patients may receive additional treatment to ensure best care.

SUMMARY:
Fever is a common symptom in many health conditions, but current methods to monitor body temperature (BT) are either invasive, costly, or not continuous. The Corsano CardioWatch 287-2, a wristband that tracks multiple vital signs, offers a new way to monitor BT by measuring skin temperature and heat flux on the wrist. It uses a machine learning algorithm to predict BT in real-time. The device has shown good results when compared to other non-invasive temperature measurements, like tympanic (ear) temperature, in stroke patients. However, it hasn't yet been compared to the gold standard of invasive rectal temperature monitoring in a clinical setting. This study aims to test the accuracy of the Corsano CardioWatch 287-2 in measuring body temperature against rectal temperature monitoring in a clinical environment.

DETAILED DESCRIPTION:
Rationale Fever is one of the most common clinical symptoms. So far, clinically established methods to monitor body temperature (BT) are either invasive and expensive (blood, bladder or rectal catheter) and/or non-continuous (tympanic temperature measurements). A continuous and scalable BT monitoring solution is missing. The Corsano CardioWatch 287-2 is a wristband intended to monitor multiple vital signs, including BT. It does so by continuously measuring the wrist's skin temperature and corresponding heat flux, from which it predicts the BT. These BT predictions are performed in real-time by a machine learning algorithm on the wearable itself. The sensor system was shown to have good correlation with tympanic temperature measurements in an acute stroke clinical setting [1]. However, a clinical validation study in which the temperature sensor of the Corsano CardioWatch 287 is compared to invasive rectal temperature monitoring, is lacking.

Research objective This study's research objective is to investigate the validity of BT measurement through skin temperature and skin heat flux measurement by the Corsano CardioWatch 287-2 against invasive rectal temperature monitoring in a clinical setting.

Primary objective The main objective is to validate the clinical accuracy of BT spot measurements by the Corsano CardioWatch 287-2 according to ISO 80601-2-56;2017+A1;2018 [1,2].

Secondary objective The secondary objective is to compare continuous BT measurements by the Corsano CardioWatch 287-2 with measurements from a clinically conventional, continuous rectal temperature sensor. Bias and limits of agreement for CardioWatch 287-2 will also be calculated in comparison to the rectal temperature probe measurements.

As a third goal, simultaneously available thermometer readings of clinical thermometers, such as Radius-T temperature readings, tympanic temperature readings and rectal temperature probe readings, will be compared with each other to assess the difference in respect to each other.

The fourth goal of this study will be to record and evaluate adverse events from the wearable BT sensor (e.g., rash).

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old;
* Able to provide consent
* Administered at the ICU or recovery room of the Reinier de Graaf hospita

Exclusion Criteria:

* Unable to wear the Corsano CardioWatch 287 or Radius-T sensor due to reasons such as allergic reactions, wounds, amputations etc.;
* Unable to receive rectal temperature monitoring;
* Thermoregulatory problems or diseases;
* Hyperthermia (>40°C);
* Known allergy to plastics / latex;
* Patient not willing to sign informed consent;
* Significant mental or cognitive impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We aim to include 120 individuals (mixed gender), of which 30-50% are displaying fever (>38°C), who are administered to the intensive care unit or the recovery room of the Reinier de Graaf Gasthuis.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Agreement between four temperature readings | From enrollment up to 24 hours
  The primary objective of this study is to compare the body temperature readings of the BT sensor with temporally corresponding tympanic thermometer, Radius-T temperature sensor and rectal thermometer readings in 120 subjects. To comply with ISO 80601-2-56;A1:2018 [1,2], the data of the four thermometers will be simplified to one temperature data point per thermometer and participant, leading to a temperature quadruplet per participant. To ensure that each subject contributes an equal proportion or weight to the total number of samples, the samples will be stratified over subjects and temperature measurement ranges. This means that the samples for each subject in each range will be upsampled by randomly selecting samples with replacement until the maximum number of samples found over all ranges and all participants is reached.
  The temperature quadruplet data points will be derived from simultaneous temperature readings taken by the four devices.
Clinical repeatability calculation | From enrollment up to 24 hours
  In order to reduce potential bias by missing temperature measurements and variability in temperature readings within individual patients the clinical repeatability will be calculated complying with ISO 80601-2-56;A1:2018 [1,2]. First, the standard deviation ,j, of the quadruplet temperature measurements for each subject j will be calculated. Subsequently, the pooled standard deviation (clinical repeatability), r, for all subjects is calculated.

SECONDARY OUTCOMES:
Agreement between temperature reading of CardioWatch 287-2 and rectal temperature probe | From enrollment up to 24 hours
  The secondary objective of this study will be to compare the continuous temperature from the CardioWatch 287-2 measurement to available continuous clinical thermometer reading, collected by the rectal temperature probe. Additionally the bias and limits of agreement for the CardioWatch 287-2 in comparison to the rectal temperature probe measurements will be calculated. For this, three measures of quality will be determined: one is the mean absolute error (MAE) between the BT prediction of the CardioWatch 287-2 and the reference signal where the mean is taken over the whole measurement of a single candidate. The other two measures of quality are the bias and 2 standard deviations.
  To investigate the third objective, the clinical bias and limits of agreement will be determined for clinical thermometer readings at the same point in time for the same participant (coming from tympanic thermometer and rectal temperature probe). This will be done according to the same method used for the pri

CONTACTS AND LOCATIONS:
Overall Officials: Mariska van Vliet, MD, PhD, Principal Investigator — Reinier de Graaf Groep
Locations (1):
- Reinier de Graaf Gasthuis, Delft, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No